CLINICAL TRIAL: NCT07056920
Title: Tomographic Evaluation of The Dimensional Changes After Horizontal Ridge Augmentation of the Lower Posterior Mandible Using a Novel Customized Porous Zirconia Shell Technique: Clinical Case Study.
Brief Title: Evaluation of Horizontal Bone Gain of Ridge Augmentation Using Customized Porous Zirconia Shell.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Shawky (Other)
Responsible Party: Sponsor-Investigator, Ahmed Shawky, Dr., October University for Modern Sciences and Arts
Organization: October University for Modern Sciences and Arts (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER 4.4.1
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Horizontal Ridge Deficiency; Deficient Alveolar Bone
Keywords: ridge augmentation; horizontal ridge augmentation; deficient alveolar ridge; zirconia; non resorbable membrane; khoury technique; zirconia membrane; lingual flap advancement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zirconia membrane (Experimental): Customized Zirconia membrane will be used as a non resorbable membrane for horizontal ridge augmentation of deficient posterior mandibular region.
  Interventions: Procedure: Zirconia shell technique

INTERVENTIONS:
Procedure: Zirconia shell technique — Customized Zirconia membrane will be printed as a porous shell and will be used as a non resorbable membrane for horizontal ridge augmentation of deficient posterior mandibular region.

SUMMARY:
Khoury technique, which employs autogenous bone blocks harvested from the patient, has been widely used for horizontal and vertical ridge augmentation. This method introduces critical limitations, including the technical complexity, morbidity associated with donor site harvesting, such as infection, neurosensory disturbances, and post-operative discomfort

This clinical case series aims to demonstrate how customized pours zirconium shell could be an alternative technique for ridge augmentation to overcome the limitations of Khoury shell technique.

DETAILED DESCRIPTION:
Ridge augmentation is a surgical procedure designed to increase the height and width of the alveolar ridge to provide adequate bone volume for the placement of dental implants. Deficient alveolar ridges are treated using various surgical techniques to restore adequate bone volume for dental implant placement. These techniques include guided bone regeneration (GBR), ridge splitting, distraction osteogenesis, autogenous block bone grafting, onlay bone grafting, and maxillary sinus lifting.

The Khoury technique is a widely recognized approach in dental implantology for horizontal and vertical ridge augmentation. This technique involves the use of autogenous bone blocks harvested from the patient, typically from the mandibular symphysis or ramus. These bone blocks are split into thin laminae and stabilized with micro screws to reconstruct deficient alveolar ridges , and the voids created between the bone blocks are filled with autogenous bone chips to promote regeneration .

This approach is associated with risks, such as donor site morbidity, infection, and potential neurosensory disturbances, sever post operative pain, also technical complexity of the procedure also restricts its application to highly skilled clinicians and patients with adequate donor sites.

These challenges highlight the need for alternative techniques or improved strategies to overcome the limitations of the Khoury technique while achieving predictable outcomes in ridge augmentation procedures.

Zirconia is utilized in the fabrication of zirconia crowns and dental implants, among other dental replacement components. This material is a polycrystalline ceramic with high strength and rigidity, even at small thickness, and bio inertness, among other interesting properties.

The structural integrity of zirconium membranes makes them an excellent choice as non-resorbable membrane for GBR. Studies have demonstrated their excellent biocompatibility, optimal tissue integration, high mechanical strength that ensured effective space maintenance for bone formation, smooth surface that minimized soft tissue ingrowth. Additionally, zirconia's customizable nature allows for precise defect contouring, leading to improved aesthetic outcomes. Overall, zirconia membranes present a valuable tool in GBR procedures, offering potential advantages over traditional materials like titanium meshes .

All those studies used the zirconia as an occlusive 3D non-resorbable membrane except on animal study evaluated the effect of the porous zirconia membrane in comparison to the occlusive one .

In an attempt to overcome the limitation of Khoury technique, zirconia can be used as a shell to augment the deficient alveolar ridges. Hence the purpose of this clinical case series is to introduce a novel customized pours zirconium shell and to tomographically assess the bone gain after horizontal ridge augmentation for deficient mandibular ridges.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* Deficient lower posterior area (Seibert class I).
* Enough inter-arch space for placement of implant-supported prosthesis.
* Motivated the patient to have the treatment.
* Good oral hygiene.

Exclusion Criteria:

* Patient with systematic conditions that could interfere with healing process.
* Pregnant females
* Smokers.
* Poor oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain | 6 months postoperatively.
  Tomographic evaluation of the horizontal bone gain using CBCT in millimeters , CBCT scans will be performed to assess the amount of bone gain in comparison to the preoperative CBCT scans

SECONDARY OUTCOMES:
Soft tissue dehiscence | Soft tissue will be evaluated post-operatively at 1, 2, 4, 6, 8, 12, and 16 week recall appointments
  Any Zirconia membrane exposure at the incision line during the healing period will be considered as soft tissue dehiscence. It will evaluated by:
  1. Clinical inspection: Yes or No
  2. any oft tissue dehiscence will be classified according to Fontana Classification (Fontana et al 2011) as:
     * Class I: Small membrane exposure (≤ 3 mm) without purulent exudate.
     * Class II: Large membrane exposure (> 3 mm) without purulent exudate.
     * Class III: Membrane exposure with purulent exudate.
     * Class IV: Abscess formation without membrane exposure.
Swelling score | Swelling score will be evaluated for one week postoperatively
  Any Swelling at the surgical area will be evaluated using the Visual Analog Scale (VAS) (0 = no swelling, 4 = extensive swelling) for 1 week postoperatively.
  The participants will be instructed to record the presence of the swelling and its degree in swelling chart as follow:
  1. No swelling
  2. Slight (Intraoral swelling at surgical site that cannot be recognized by others)
  3. Moderate (Intraoral swelling at surgical site that can be recognized by others)
  4. Extensive (Extra-oral swelling that extends beyond surgical site)
Pain score | First thing in the morning for the first 7 days post-operatively.
  Pain intensity will be evaluated using the Numerical Rating Scale (NRS) (0 = no pain, 10 = worst pain imaginable). Patients will record the pain score in the pain chart that will be collected at week 1 recall appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R Abd Elrahman, Professor, Study Director — Modern Science and Arts University; Nada Zazou, Lecturer, Study Chair — Modern Science and Arts University; Ahmed S Refaey, Bachelor, Principal Investigator — Modern Science and Arts University; Rasha Attia, Lecturer, Study Chair
Locations (1):
- October University for modern sciences and arts (MSA University), Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Study results will be shared via publication in dental journal.